CLINICAL TRIAL: NCT01302392
Title: A Randomized, Open-label, Phase 3 Study of Carfilzomib vs Best Supportive Care in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of Carfilzomib vs Best Supportive Care in Subjects With Relapsed and Refractory Multiple Myeloma
Acronym: FOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-011
Record Dates: First submitted 2011-02-10; First posted 2011-02-24 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best Supportive Care (Active Comparator)
  Interventions: Drug: Best Supportive Care
- Carfilzomib (Experimental)
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — 20mg/m² IV on Days 1 and 2 of Cycle 1, escalating to 27 mg/m² IV on Days 8,9,15,and 16 of Cycle 1 and continuing on Days 1,2,8,9,15,and 16 of Cycles 2 through Cycle 9. Cycles 10 and beyond will receive 27 mg/m² IV on Days 1,2,15, and 16 (alternatively, the investigator could choose to continue the dosing frequency on the original dosing days [Days 1, 2, 8, 9, 15, 16] for individual subjects).
  Other Names: PR-171
  Arms: Carfilzomib
Drug: Best Supportive Care — Corticosteroid (either prednisolone 30 mg orally (PO) every other day, dexamethasone 6 mg PO every other day, or other equivalent corticosteroid).
  Optional cyclophosphamide 50 mg PO once daily may be given at the Investigator's discretion (maximum of 1400 mg per 28-day cycle).
  Arms: Best Supportive Care

SUMMARY:
This is a Phase 3, randomized, open-label, multicenter study comparing two treatment regimens for subjects with multiple myeloma who have received all available approved treatment options and may therefore be considered candidates for palliative care.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma
2. Measurable disease based on central laboratory values, as defined by one or both of the following criteria (assessed within 21 days prior to randomization):

   * Serum M-protein

     * Serum protein electrophoresis (SPEP): ≥ 0.5 g/dL
     * For immunoglobulin A (IgA) patients whose disease can only be reliably measured by serum quantitative immunoglobulin (qIgA): > 750 mg/dL (0.75 g/dL)
   * Urine Bence Jones protein: ≥ 200 mg/24 h
3. Responsive (defined as a 25% or greater decrease in M-protein or total protein) to at least one line of prior therapy
4. Relapsed multiple myeloma, defined as disease progression while on or after at least 1 prior treatment regimen
5. Refractory multiple myeloma, defined as meeting one or more of the following:

   * Nonresponsive to most recent therapy (eg, stable disease only, or progressive disease while on treatment)
   * Disease progression within 60 days of discontinuation from most recent therapy
6. Received 3 or more prior therapeutic regimens for multiple myeloma
7. Adequate prior treatment with bortezomib (if less than 4 complete cycles, the reason for discontinuation must be reviewed by the Medical Monitor and the reason documented)
8. Prior treatment with an immunomodulatory agent (lenalidomide, if available, and/or thalidomide)
9. Prior treatment with an alkylating agent (standard or high-dose)
10. Prior treatment with a corticosteroid
11. Criterion no longer applicable (with Amendment 2, Criterion 11, the requirement of "prior treatment with an anthracycline unless not clinically indicated" is removed.)
12. Age ≥ 18 years
13. Life expectancy of at least 1 month
14. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
15. Adequate hepatic function, with serum alanine aminotransferase (ALT) < 4 times the upper limit of normal and serum bilirubin < 2.5 mg/dL (42.5 µmol/L). Patients with total bilirubin ≥ 2.5 mg/dL may enrol if their serum direct bilirubin is < 2.5 mg/dL.
16. Total white blood cell (WBC) count ≥ 1.5 × 10^9/L and absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L (use of colony-stimulating factors to achieve these counts is allowed)
17. Hemoglobin ≥ 7.5 g/dL (75 g/L)

    -Use of erythropoietic stimulating factors is allowed:
    * For all patients who receive a red blood cell (RBC) transfusion within 28 days of obtaining the Screening hemoglobin value. The following information must be provided for the Medical Monitor's review for assessment for eligibility:

      * Pre-transfusion hemoglobin (Hb)
      * Number of RBC units administered
      * Use of erythropoietic stimulating factors
18. Platelet count ≥ 30 × 10^9/L

    -There is no restriction on platelet transfusions or thrombopoietic growth factor before or during the screening period
    * For all patients who receive a platelet transfusion within 7 days of obtaining the Screening platelet value, the following information must be provided for the Medical Monitor's review for assessment of eligibility

      * Pre-transfusion platelet count
      * Number of platelet units administered
      * Use of thrombopoietic growth factors
19. Creatinine clearance (CrCl) ≥ 15 mL/minute (either measured or calculated using a standard formula such as Cockcroft and Gault) and dialysis-independent
20. Written informed consent in accordance with regulatory guidelines
21. Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of the first dose of study treatment and agree to use an effective method of contraception during the study and for 3 months following the last dose of study treatment. Post-menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential.

Exclusion Criteria:

1. Waldenström's macroglobulinemia or IgM myeloma
2. Refractory to all prior therapies
3. Disease measurable only by serum free light chain assay (SFLC)
4. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
5. Plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
6. Prior carfilzomib treatment
7. Chemotherapy (approved or investigational) within 14 days prior to randomization
8. Immunotherapy or antibody therapy within 28 days prior to randomization
9. Corticosteroid therapy at a dose equivalent to dexamethasone > 4 mg/day within 14 days prior to randomization
10. Radiotherapy within 7 days prior to randomization
11. Major surgery within 21 days prior to randomization
12. Congestive heart failure (NYHA Class III or IV) or symptomatic cardiac ischemia, conduction system abnormalities uncontrolled by conventional intervention (conduction abnormalities not clinically warranting intervention are allowed)
13. Myocardial infarction in the previous 3 months
14. Acute active infection requiring systemic treatment (antibiotics, antivirals, or antifungals) within 14 days prior to randomization
15. Known human immunodeficiency virus seropositivity
16. Active hepatitis A, B, or C infection
17. Other malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix, vulva, or breast; c) prostate cancer of Gleason Score 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder, carcinoma in situ of the breast, or benign tumors of the adrenal or pancreas
18. Significant neuropathy (Grades 3-4, or Grade 2 with pain) at the time of randomization
19. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent
20. Pregnant or lactating females
21. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity or known history of allergy to carfilzomib, Captisol® (a cyclodextrin derivative used to solubilize carfilzomib) all anticoagulation and antiplatelet options, antiviral drugs; or intolerance to hydration due to preexisting pulmonary or cardiac impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2010-09; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (68):
- Australia (2):
  - Nedlands
  - Perth
- Austria (3):
  - Linz
  - Salzburg
  - Vienna
- Belgium (4):
  - Arlon
  - Bruges
  - Brussels
  - Roeselare
- Czechia (4):
  - Brno
  - Hradec Kralov
  - Olomouc
  - Prague
- France (3):
  - Lyon
  - Nantes
  - Nîmes
- Germany (6):
  - Dresden
  - Giessen
  - Koblenz
  - Mainz
  - München
  - Ulm
- Greece (2):
  - Athens
  - Rio Patras
- Hungary (7):
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Pécs
  - Szeged
- Israel (6):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nahariva
  - Petah Tikva
  - Sheba
- Italy (4):
  - Ancona
  - Novara
  - Roma
  - Torino
- North Shore, New Zealand
- Poland (7):
  - Gdansk
  - Lodz
  - Piła
  - Torum
  - Warsaw
  - Wroclaw
  - Zamość
- Russia (2):
  - Moscow
  - Saint Petersburg
- Serbia (2):
  - Belgrade
  - Niš
- Bratislava, Slovakia
- South Korea (2):
  - Incheon
  - Seoul
- Spain (7):
  - Barcelona
  - Guipuzcoa
  - Murcia
  - Salamanca
  - Seville
  - Valencia
  - Zaragoza
- Uppsala, Sweden
- United Kingdom (4):
  - Hampshire
  - London
  - Manchester
  - Oxford

REFERENCES:
- [Derived] Hajek R, Masszi T, Petrucci MT, Palumbo A, Rosinol L, Nagler A, Yong KL, Oriol A, Minarik J, Pour L, Dimopoulos MA, Maisnar V, Rossi D, Kasparu H, Van Droogenbroeck J, Yehuda DB, Hardan I, Jenner M, Calbecka M, David M, de la Rubia J, Drach J, Gasztonyi Z, Gornik S, Leleu X, Munder M, Offidani M, Zojer N, Rajangam K, Chang YL, San-Miguel JF, Ludwig H. A randomized phase III study of carfilzomib vs low-dose corticosteroids with optional cyclophosphamide in relapsed and refractory multiple myeloma (FOCUS). Leukemia. 2017 Jan;31(1):107-114. doi: 10.1038/leu.2016.176. Epub 2016 Jun 24. PMID 27416912
- [Derived] Hajek R, Bryce R, Ro S, Klencke B, Ludwig H. Design and rationale of FOCUS (PX-171-011): a randomized, open-label, phase 3 study of carfilzomib versus best supportive care regimen in patients with relapsed and refractory multiple myeloma (R/R MM). BMC Cancer. 2012 Sep 19;12:415. doi: 10.1186/1471-2407-12-415. PMID 22992303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 06 Sep 2010 to 21OCT2012. Results are reported as of the data cut-off date of 10 Jul 2014.
Period: Overall Study
Arm/Group | Best Supportive Care | Carfilzomib
Started | 158 | 157
Treated | 153 | 157
Completed | 151 | 156
Not Completed | 7 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Best Supportive Care | Carfilzomib | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.02) | 63.3 (10.71) | 64.4 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 75 | 137
  Male | 96 | 82 | 178
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 148 | 151 | 299
  Other | 5 | 4 | 9
Region [Number; unit: participants]
  Europe | 138 | 140 | 278
  Non-Europe | 20 | 17 | 37
Number of Prior Regimens to Treat Multiple Myeloma [Number; unit: participants]
  3 | 19 | 17 | 36
  4 | 35 | 34 | 69
  ≥5 | 104 | 106 | 210

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time elapsed between the randomization date and the date of death. Participants who were still alive were censored at date when the subject is last known alive or the data cutoff date, whichever occurs earlier.
Time Frame: From randomization through the final analysis data cutoff with longest follow-up time of approximately 45 months. Median follow up times were 27.8 months and 29.8 months for Carfilzomib and Best Supportive Care groups, respectively.
Population: The intent to treat (ITT) analysis set comprised all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 158 | 157
months | 10.0 [7.7 to 12.0] | 10.2 [8.4 to 14.4]
Statistical Analysis 1: Comparison: Best Supportive Care vs Carfilzomib; Test type: Superiority or Other; p = 0.4172, Log Rank — Based on 1-sided test; Analysis was stratified by the number of previous therapies (3 vs 4 vs ≥ 5) and geographical region (Europe vs. non-Europe); Hazard Ratio (HR) = 0.975, 95% CI 2-sided [0.760 to 1.249]

2. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier estimate of median time from randomization to progressive disease (PD) or all-cause death. PD was assessed using International Myeloma Working Group-Uniform Response Criteria (IMWG-URC). 1 or more conditions were required to meet PD: 2 consecutive rising serum or urine M-protein from central lab; documented new bone lesion(s) or soft tissue plasmacytoma(s) or increased size of existing bone lesion(s) or plasmacytoma(s); or confirmed hypercalcemia due solely to plasma cell proliferative disorder (local lab greater than 11.5 mg/dL on 2 separate occasions). Censoring conditions (censoring dates) were: no post-baseline disease assessment (DA) (randomization date); started non-protocol systemic anticancer treatment before PD or death (last DA date before such treatment); died or had PD after more than 1 missed DA (last DA date without PD before the first missed visit); or were alive and without documentation of PD, including lost to follow-up without PD (last DA date).
Time Frame: From randomization through the final analysis data cutoff with longest follow-up time of approximately 31 months. Median follow up times were 26.6 months and 23.1 months for Carfilzomib and Best Supportive Care groups, respectively.
Population: The intent to treat (ITT) analysis set comprised all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 158 | 157
months | 3.3 [2.2 to 5.2] | 3.7 [2.8 to 4.2]

3. Secondary Outcome: Overall Response
Description: Number of participants who achieved confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) as their best response. Response was determined using the International Myeloma Working Group - Uniform Response Criteria (IMWG-URC).
Time Frame: as for outcome 2
Population: The intent to treat (ITT) analysis set comprised all randomized participants.
Measure: Number; unit: participants
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 158 | 157
participants | 18 | 30

4. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was calculated for subjects who achieved a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR). Duration of response was defined as the time in months from the initial start of response (PR or better) to the earlier of documented progressive disease (PD) or death due to any cause. Participants who had not progressed or died were censored according to the censoring rules defined previously for progression-free survival.
Time Frame: From the time achieving response through the final analysis data cutoff with longest follow-up time of approximately 29 months.
Population: The intent to treat (ITT) population comprised randomized participants who achieved a best overall response of PR or better only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 18 | 30
months | 9.5 [3.7 to NA] — Upper limit of the confidence interval not calculable due to a low number of participants reaching PD or all-cause death. | 7.2 [4.6 to 12.0]

5. Secondary Outcome: Clinical Benefit Response
Description: Number of participants who achieved confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), or minimal response (MR) as their best response. Response was determined using the International Myeloma Working Group - Uniform Response Criteria (IMWG-URC). (MR was determined using European Group for Blood and Marrow Transplantation criteria)
Time Frame: as for outcome 2
Population: The intent to treat (ITT) analysis set comprised all randomized participants.
Measure: Number; unit: participants
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 158 | 157
participants | 33 | 49

6. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of Clinical Benefit was calculated for subjects who achieved a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR) or minimal response (MR). Duration of Clinical Benefit was defined as the time in months from the initial start of response (MR or better) to the earlier of documented progressive disease (PD) or death due to any cause. Participants who had not progressed or died were censored according to the censoring rules defined previously for progression-free survival.
Time Frame: From time of achieving clinical benefit through the final analysis data cutoff with longest follow-up time of approximately 30 months.
Population: The intent to treat (ITT) population comprised randomized participants who achieved a best overall response of MR or better only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 33 | 49
months | 8.3 [6.5 to 12.9] | 6.4 [4.9 to 8.3]

7. Secondary Outcome: Disease Control
Description: Number of participants who achieved confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal response (MR), or stable disease (SD) lasting ≥ 8 weeks as their best response. Response was determined using the International Myeloma Working Group - Uniform Response Criteria (IMWG-URC). (MR was determined using European Group for Blood and Marrow Transplantation criteria)
Time Frame: as for outcome 2
Population: The intent to treat (ITT) analysis set comprised all randomized participants.
Measure: Number; unit: participants
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 158 | 157
participants | 107 | 119

8. Secondary Outcome: Duration of Disease Control
Description: Duration of Disease Control was calculated for subjects who achieved disease control. Duration of Disease Control was defined as the time in months from randomization to the earlier of documented progressive disease (PD) or death due to any cause. Participants who had not progressed or died were censored according to the censoring rules defined previously for progression-free survival.
Time Frame: From time of achieving disease control through the final analysis data cutoff with longest follow-up time of approximately 31 months.
Population: The intent to treat (ITT) population comprised randomized participants who achieved disease control.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Best Supportive Care | Carfilzomib
Number analyzed (Participants) | 107 | 119
months | 6.6 [5.4 to 8.8] | 5.5 [3.9 to 6.5]

ADVERSE EVENTS:
Time Frame: From randomization through the final analysis data cutoff with range of follow-up time of 0.4 - 138.3 weeks with median of 10.7 weeks in Best Supportive Care arm, and 0.3 - 138.4 weeks with median of 16.3 weeks in carfilzomib arm
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Best Supportive Care | Carfilzomib
Serious Adverse Events (participants affected / at risk) | 78/153 | 92/157
Other Adverse Events (participants affected / at risk) | 135/153 | 141/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Best Supportive Care (N=153) | Carfilzomib (N=157)
Anaemia (Blood and lymphatic system disorders) | 8 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 1 | 4
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 19 | 16
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 6
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 3
Bronchopneumonia (Infections and infestations) | 5 | 6
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 18 | 10
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 1 | 3
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 3 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Renal failure acute (Renal and urinary disorders) | 6 | 15
Renal impairment (Renal and urinary disorders) | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Best Supportive Care (N=153) | Carfilzomib (N=157)
Anaemia (Blood and lymphatic system disorders) | 72 | 88
Leukopenia (Blood and lymphatic system disorders) | 15 | 9
Neutropenia (Blood and lymphatic system disorders) | 23 | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 43 | 58
Constipation (Gastrointestinal disorders) | 20 | 10
Diarrhoea (Gastrointestinal disorders) | 18 | 23
Dyspepsia (Gastrointestinal disorders) | 4 | 10
Nausea (Gastrointestinal disorders) | 14 | 31
Vomiting (Gastrointestinal disorders) | 5 | 15
Asthenia (General disorders) | 20 | 26
Chest pain (General disorders) | 8 | 5
Chills (General disorders) | 1 | 8
Fatigue (General disorders) | 28 | 29
Oedema peripheral (General disorders) | 12 | 17
Pain (General disorders) | 1 | 8
Pyrexia (General disorders) | 28 | 41
Bronchitis (Infections and infestations) | 13 | 13
Nasopharyngitis (Infections and infestations) | 10 | 13
Respiratory tract infection (Infections and infestations) | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 3 | 16
Blood creatinine increased (Investigations) | 10 | 13
Creatinine renal clearance decreased (Investigations) | 4 | 9
Neutrophil count decreased (Investigations) | 10 | 13
Platelet count decreased (Investigations) | 12 | 12
Decreased appetite (Metabolism and nutrition disorders) | 7 | 9
Hypercalcaemia (Metabolism and nutrition disorders) | 9 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 8
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 19
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 16 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 13
Dizziness (Nervous system disorders) | 3 | 10
Headache (Nervous system disorders) | 6 | 17
Insomnia (Psychiatric disorders) | 18 | 4
Renal failure (Renal and urinary disorders) | 3 | 8
Renal impairment (Renal and urinary disorders) | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Hypertension (Vascular disorders) | 9 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.